CLINICAL TRIAL: NCT06711146
Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10-19) in the Treatment of Moderate to Severe Active SLE Clinical Research
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meta10-19-007
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Meta10-19; CAR-T Cells Therapy; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of Metabolically Armed CD19 CAR-T cells (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion. A dose of metabolically armed CD19 CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed CD19 CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed CD19 CAR-T cells — Each subject receive metabolically armed CD19 CAR- T cells by intravenous infusion
  Other Names: Meta10-19

SUMMARY:
A Study of Metabolically Armed CD19 CAR-T Cells Therapy for Patients With Moderate to Severe Active Systemic Lupus Erythematosus

DETAILED DESCRIPTION:
This is a single arm, open-label study. This study is indicated for moderate to severe active systemic lupus erythematosus. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products and our earlier disclosed clinical trials .

1. Main research objectives:

   To evaluate the safety and efficacy of metabolically armed CD19 CAR-T Cells in the treatment of moderate to severe active SLE.
2. Secondary research objectives:

(1) To evaluate the pharmacokinetic (PK) and pharmacodynamics(PD) characteristics of metabolically armed CD19 CAR-T Cells after infusion and their relationship with the number of B cells.

(2) To evaluate the effects of the concentration of autoimmune antibodies and complement after infusion of metabolically armed CD19 CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

* All subjects or guardians must sign an informed consent form approved by the Ethics Committee in person before commencing any screening process;
* Be over 18 years of age, male or female;
* A diagnosis of SLE according to the 2012 systemic lupus international collaborating clinics(SLICC);
* The history of SLE prior to screening was at least 6 months, and the disease remained active at least 2 months after the use of a stable standard SLE regimen prior to screening:

  1. Conventional regimens for SLE are corticosteroids and one or more immunomodulatory drugs over 6 months；
  2. Oral corticosteroids must meet the following requirements:

     * Prednisone (or equivalent) ≥7.5 mg/ day, and ≤60 mg/ day；
     * There is no minimum daily dose requirement for corticosteroids when used in combination with immunosuppressants；
     * At least 8 weeks of treatment prior to screening, and the dose must be kept stable for > 2 weeks.
* Screening is positive for antinuclear antibodies, and/or anti-DS-DNA antibodies, and/or anti-Smith antibodies；
* SELENA-SLEDAI score ≥8 during the screening period. Score ≥6 for SELENA-SLEDAI clinical symptoms (except for low complement and/or anti-DS-DNA antibodies) if low complement and/or anti-DS-DNA antibody score is present；
* Women of childbearing age and all male patients must consent to use a effective contraception for at least 12 months after Meta10-19 infusion and until two consecutive PCR tests show no more CAR T cells in vivo;
* CD19 expression was positive by or flow cytometry ;
* Organ function：

  1. Complete blood count (CBC) test [the following criteria should be met within 24 hours prior to apheresis, and supportive treatment such as transfusion, platelet transfusion, cell growth factor (except recombinant erythropoietin) should be avoided within 7 days prior to detection]

     * Lymphocyte count ≥ 0.5×109/L (except for those receiving bridging chemotherapy);
     * Platelet count ≥ 25×109/L;
     * Hemoglobin ≥ 70.0 g/L
  2. Blood Biochemistry:

     * Serum creatinine (Scr) ≤ 1.5 x ULN, or
     * endogenous creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault formula);
     * alanine aminotransferase (ALT) ≤ 2.5 x ULN;
     * aspartate aminotransferase (AST) ≤ 2.5 ×ULN;
     * Total bilirubin (TBIL) ≤ 2 ×ULN; Subjects with total bilirubin < 3 × ULN and direct bilirubin < 1.5× ULN with Gilbert-.Meulengracht syndrome could be included;
     * Serum lipase and amylase ≤ 1.5×ULN;
     * Alkaline phosphatase (ALP) ≤ 2.5 ×ULN;
     * In case of bone or liver metastasis, AST, ALT and ALP ≤ 5 ×ULN;
     * Prothrombin time (PT) extended ≤ 4 s, fibrinogen ≥ 1 g/L, activated partial thromboplastin time (APTT) ≤ 1.5 ×ULN;
  3. Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) > 91% in indoor air environment..
* Hemodynamic stability was determined by echocardiography or multichannel radionuclide angiography (MUGA) and LVEF ≥45％.

Exclusion Criteria:

* Severe lupus nephritis (defined as proteinuria > 6 g/24h or serum creatinine > 2.5 mg/dL or 221 μmol/L), treatment with active nephritis with Prohibited drugs, hemodialysis, or prednisone ≥100 within 8 weeks prior to screening mg/d or equivalent glucocorticoid therapy ≥14 days.
* Prior to screening, other lupus crises, such as active central nervous system lupus, severe hemolytic anemia, severe thrombocytopenic purpura, severe agranulocytosis, severe myocardial damage, severe lupus pneumonia or pulmonary hemorrhage, severe lupus hepatitis, and severe vasculitis.
* Clinically significant central nervous system diseases or pathological changes not caused by lupus prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
* Combined with other autoimmune diseases, systematic treatment is needed.
* History of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
* IgA deficiency was present during screening (serum IgA level < 10 mg/dL).
* Other conditions that the investigator considered should not be enrolled in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 35 days of study treatment.
  Determine the Maximal Tolerable Dose(MTD).
DCR | 3 and 6 months following infusion of Meta10-19.
  Disease control rates (DCR) assessed according to SLEDAI-2000, Physician Overall Assessment (PGA), and medication.

SECONDARY OUTCOMES:
Concentration of CAR-T cells | Up to 12 months after CAR-T treatment.
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion.
Pharmacodynamics of CAR-T cells | Up to 28 days after infusion.
  Concentration levels of CAR-T related serum cytokines such as CRP, IL-6, INF-γ at each time point.
Autoantibody detection | Up to 12 months after CAR-T treatment
  Concentration levels of B cell related serum antibodies such as complement factor C3 , ANA, anti-dsDNA each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No